CLINICAL TRIAL: NCT02331186
Title: Effects of Bariatric Surgery on Pelvic Floor in Obese Women
Brief Title: Effects of Bariatric Surgery on Pelvic Floor Fonctions in Obese Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Hediye Dagdeviren, M.D., Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2014/11/01
Record Dates: First submitted 2014-12-21; First posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Urinary Incontinence; Obesity
Keywords: Obesity; Bariatric surgery; Urinary incontinence; Pelvic floor
MeSH Terms: conditions — Urinary Incontinence; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obese women who underwent bariatric surgery: obese women who underwent bariatric surgery
  Interventions: Procedure: bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgery — bariatric surgery for obese women

SUMMARY:
Urinary incontinence is well documented as a comorbidity of obesity. Studies demonstrate improvement of incontinency after weight loss. However, the mechanisms are still not clear. Aim of our study to analyze the effects of bariatric surgery on pelvic floor function in women.

DETAILED DESCRIPTION:
Obesity is considered an important public health problem, both in developed and developing countries. Obese people are at a higher risk for developing various comorbidities: type II diabetes, dyslipidemia, cardiovascular and cerebrovascular diseases, coagulation disorders, degenerative joint disease, some types of cancer, sleep apnea and urinary incontinence Women suffering from obesity are more likely to develop urinary incontinence, especially when related to stress. Excess weight is a modifiable risk factor. It is believed that weight reduction may be an effective treatment for urinary incontinence. The aim of this study is to analyze the effects of weight loss induced by bariatric surgery on pelvic floor function. Taking into account that modest weight loss (5% to 10%) already brings benefits to women with obesity and incontinence, one may assume even more marked improvement owing to the massive loss of weight by surgical means.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 40 kg/m2
* >18 years old
* participants who provided written informed consent

Exclusion Criteria:

* History of gynecologic operation time under one year
* History of pelvic physiotherapy
* Chronic obstructif lung disease
* Norologic disease
* Women in menopause

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women who underwent bariatric surgery Body mass index ≥ 40 kg/m2 >18 years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
urodynamic parameters | after six month
  effect of bariatric surgery on urodynamic parameters in obese women

SECONDARY OUTCOMES:
Urinary incontinence | after six month
  effect of bariatric surgery on urinary incontinance in obese women
oxford scales | after six month
  effect of bariatric surgery on oxford scales in obese women
health quality scores | after six month
  effect of bariatric surgery on health quality scores in obese women

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Bakirkoy Dr Sadi Konuk Training and Research Hospital, Istanbul, Bakirkoy
  - Bakirkoy Dr. Sadi Konuk Teaching and Research Hospital, Istanbul, Istanbul